CLINICAL TRIAL: NCT02641561
Title: Prevention of Post-Endoscopic Retrograde Cholangiopancreatography (ERCP) - Induced Pancreatitis Using Aggressive Lactated Ringer's Infusion and/or Rectal Indomethacin
Brief Title: Lactated Ringers With or Without Rectal Indomethacin to Prevent Post-ERCP Pancreatitis
Acronym: IND+LRPEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Cooper Health System (Other)
Responsible Party: Principal Investigator, Shaffer R S Mok, Clinical Instructor, The Cooper Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 14-091
Record Dates: First submitted 2015-11-05; First posted 2015-12-29 (Estimated); Results first posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-01

CONDITIONS: Post-ERCP Acute Pancreatitis
Keywords: Pancreatitis; ERCP; Indomethacin; Lactated ringer's
MeSH Terms: conditions — Pancreatitis | interventions — Indomethacin; Ringer's Lactate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (NS+Placebo) (Placebo Comparator): Normal Saline (intravenous during procedure) + Placebo (100mg suppository per rectum prior to procedure )
  Interventions: Drug: Normal Saline; Drug: Placebo
- B (NS+IND) (Active Comparator): Normal Saline (intravenous during procedure) + Indomethacin (100mg suppository per rectum prior to procedure )
  Interventions: Drug: Indomethacin; Drug: Normal Saline
- C (LR+Placebo) (Active Comparator): Lactated ringer's solution (1 Liter, intravenous prior to procedure) + Placebo (100mg suppository per rectum prior to procedure)
  Interventions: Drug: Lactated Ringer's Solution; Drug: Placebo
- D (LR+IND) (Experimental): Lactated ringer's solution (1 Liter, intravenous prior to procedure) + Indomethacin (100mg suppository per rectum prior to procedure)
  Interventions: Drug: Indomethacin; Drug: Lactated Ringer's Solution

INTERVENTIONS:
Drug: Indomethacin — Indomethacin is a non-steroidal anti-inflammatory drug (NSAID) which is commonly used to reduce inflammation caused by gout, osteoarthritis and rheumatoid arthritis. It acts by blocking the cyclo-oxygenase 1 and 2 (COX) receptors. It has also been implicated to prevent post-ERCP pancreatitis
  Other Names: IND
  Arms: B (NS+IND); D (LR+IND)
Drug: Lactated Ringer's Solution — Lactated ringer's solution (LR), is an intravenous fluid (IVF) used commonly during endoscopic procedures and operative procedures. It's composition is similar to that of humans including sodium, chloride, potassium, calcium and lactate. Studies have implicated the use of this fluid in pancreatitis treatment and prevention of post-ERCP pancreatitis
  Other Names: LR
  Arms: C (LR+Placebo); D (LR+IND)
Drug: Normal Saline — standard IVF would include 0.9% normal saline (NS) solution used during all endoscopic procedures. 0.9% NS includes equal parts sodium and chloride.
  Other Names: NS
  Arms: A (NS+Placebo); B (NS+IND)
Drug: Placebo — Placebo would be a suppository 50 mg x 2
  Arms: A (NS+Placebo); C (LR+Placebo)

SUMMARY:
Post-ERCP pancreatitis is a well-known and sometimes life-threatening complication of ERCP. Both LR and rectal indomethacin have shown benefit in preventing post-ERCP pancreatitis. Despite this, no study to date has evaluated both of these measures for preventing post-ERCP pancreatitis. It is our hope to evaluate the combination of these two modalities for preventing post-ERCP pancreatitis compared with either modality alone.

DETAILED DESCRIPTION:
Endoscopic retrograde cholangiopancreatography (ERCP) is commonly used diagnostic and therapeutic intervention used in Gastroenterology. At Cooper University Hospital (CUH), we perform approximately 700 ERCPs per year. A known complication of ERCP is post-ERCP pancreatitis. The incidence of post-ERCP pancreatitis has been cited at anywhere from 2.6-3.5% of cases. Also, severe acute pancreatitis has been cited at rates of 0.32-0.4% and death 0.11%.

Recent literature has cited the use of several modalities useful in preventing post-ERCP pancreatitis. Among the modalities evaluated non-steroidal anti-inflammatory drugs (NSAIDS), specifically rectal indomethacin, have demonstrated benefit in preventing post-ERCP. In particular Elmunzer et al demonstrated a benefit in those with sphincter of oddi dysfunction (SOD) and those deemed "high risk" for post-ERCP pancreatitis. Other medication such at octreotoide and corticosteroid have shown mixed results.

Additionally, recent studies have demonstrated the use of lactated ringer's solution (LR) in lieu of normal saline (NS) in patient's with acute pancreatitis. Due to this thought process a recent study evaluated the use of LR in preventing post-ERCP pancreatitis. The results of this study showed that no patients who received aggressive LR hydration developed post-ERCP pancreatitis.

As rectal indomethacin and LR infusion appear to have the most definitive evidence for preventing post-ERCP pancreatitis, it is our hope to evaluate the combination of these two therapies for the prevention of post-ERCP pancreatitis.

This is a double blinded, randomized prospective cohort study involving 4 treatment groups undergoing ERCP.

All treatment arms shall receive consent, pre-procedural risk stratification, demographic data and pre-procedural liker pain scale. All subjects shall receive a study subject number and undergo randomization. All subjects also will receive post-procedural likert pain scale assessment, day 1 and 30 questioning. Treatment arms shall be separated into whether subjects are high risk or not defined in.

Time 0 (Visit 1):

Subjects undergo standard pre-procedural evaluation by nursing, anesthesia and consent for procedure/anesthesia.

The subject shall then be evaluated for study participation and subsequently consented if they desire to be part of the study. They may also undergo informed consent prior to the day of their procedure during their normal office visit. All subjects must have Liver function tests (LFTs), amylase and lipase levels drawn prior to their ERCP test. Subjects will be excluded from study participation if they have acute pancreatitis defined as;

The diagnosis of AP is most often established by the presence of 2 of the 3 following criteria:

(i) abdominal pain consistent with the disease (ii) serum amylase and / or lipase greater than three times the upper limit of normal, and / or (iii) characteristic findings from abdominal imaging

The day of their procedure, nursing shall then obtain intravenous peripheral access (standard for ERCP). Initial demographic data and risk factor data shall be obtained. Subjects shall then be randomized to one of the four study arms and given a study number randomly generated:

Pending which treatment arm the patient is enrolled into the subject shall then receive the above listed therapies and undergo their procedure.

Post-procedure the interventions performed during the ERCP shall be recorded and the patient will go through the standard recovery process. Post-procedure after recovery from anesthesia, the patients shall then be evaluated for the presence of pain after ERCP testing on the standard likert pain scale.

If the subject's pain has substantially increased from baseline, subjects shall then be admitted to the hospital and LFTs, a lipase and amylase level shall be drawn and abdominal imaging ordered if needed by the admitting physician (all the standard of care).

Time 1 Days (Visit 2 via phone):

Subjects shall be called 24 hours from ERCP to assess;

1. Presence/absence of pain
2. If pain, the severity
3. Performance of amylase and lipase
4. Whether admission, urgent care or emergency department visit did occur

Time 1-30 Days The investigator will await the subjects laboratory values and if > 3 times the upper limit of normal contact the subject via phone.

Time 30 Days (Visit 3 via phone):

Subjects shall be contacted via phone 30 days from ERCP to assess;

1. Presence/absence of pain
2. If pain, the severity
3. Whether admission, urgent care or Emergency Department (ED) visit did occur to a healthcare facility
4. Study summary

To detect a difference of 0.24 vs 0.05 a minimum of 48 per group would be needed (using p=0.05).

Descriptive statistics will be used to summarize demographic variables such as age, gender, race, length of stay, as well diagnosis and disease characteristics such as reasons for ERCP, disease intervention, pain,and outcome variables. Data tables will be generated for those variables with means, standard deviation (SD), medians, interquartile range (IQR), and confidence interval (CI). The Chi-Square test will be used to determine the main effect of treatment on ERCP induced pancreatitis. Nonparametric tests will be used to analyze categorical data while normally distributed data will be analyzed using ANOVA to look for treatment effect on other variables of interest.

Binary and Multinomial Logistic Regression will be used to examine predictors of outcome within treatments and across treatments by building interactions into the model (e.g. reasons for ERCP, intervention type). Data analysis will be performed using Systat version 13 and SPSS version 22. A p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1 Subjects who are undergoing endoscopic retrograde cholangiopancreatography (ERCP)

* Age > 18 years
* Non-pregnant
* Non-prisoners
* Subjects who can sign informed consent
* Serum Creatinine < 1.2 milligrams/deciliter (mg/dL)
* Subjects without renal failure (acute or chronic)
* Subjects without congestive heart failure (ejection fraction < 40%)
* Subjects without cirrhosis of the liver
* Subjects without allergy to aspirin or non-steroidal anti-inflammatory drugs (NSAIDS)
* Subjects not on non-steroidal anti-inflammatory drugs NSAIDS prior to enrollment

Exclusion Criteria:

* Subjects who are not undergoing ERCP
* Age < 18 years
* Pregnancy
* Prisoners
* Subjects lacking the capacity to consent for themselves
* Serum Creatinine > 1.2 milligrams/deciliter (mg/dL)
* Subjects with renal failure (acute and chronic)
* Subjects with congestive heart failure (ejection fraction < 40%)
* Subjects with cirrhosis of the liver
* Subjects with allergy to aspirin or non-steroidal anti-inflammatory drugs (NSAIDS)
* Subjects with gastrointestinal hemorrhage
* Subjects on chronic non-steroidal anti-inflammatory drugs NSAIDS
* Subjects with acute pancreatitis the day of their procedure (CITE 1-3)(APPENDIX 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaffer RS Mok, MD, MBS, Principal Investigator — The Cooper Health System
Locations (1):
- Cooper Hospital, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cotton PB, Lehman G, Vennes J, Geenen JE, Russell RC, Meyers WC, Liguory C, Nickl N. Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc. 1991 May-Jun;37(3):383-93. doi: 10.1016/s0016-5107(91)70740-2. PMID 2070995
- [Background] ASGE Standards of Practice Committee; Anderson MA, Fisher L, Jain R, Evans JA, Appalaneni V, Ben-Menachem T, Cash BD, Decker GA, Early DS, Fanelli RD, Fisher DA, Fukami N, Hwang JH, Ikenberry SO, Jue TL, Khan KM, Krinsky ML, Malpas PM, Maple JT, Sharaf RN, Shergill AK, Dominitz JA. Complications of ERCP. Gastrointest Endosc. 2012 Mar;75(3):467-73. doi: 10.1016/j.gie.2011.07.010. No abstract available. PMID 22341094
- [Background] Petersen BT. ERCP outcomes: defining the operators, experience, and environments. Gastrointest Endosc. 2002 Jun;55(7):953-8. doi: 10.1067/mge.2002.123622. No abstract available. PMID 12024166
- [Background] Tenner S, Baillie J, DeWitt J, Vege SS; American College of Gastroenterology. American College of Gastroenterology guideline: management of acute pancreatitis. Am J Gastroenterol. 2013 Sep;108(9):1400-15; 1416. doi: 10.1038/ajg.2013.218. Epub 2013 Jul 30. PMID 23896955
- [Background] Andriulli A, Loperfido S, Napolitano G, Niro G, Valvano MR, Spirito F, Pilotto A, Forlano R. Incidence rates of post-ERCP complications: a systematic survey of prospective studies. Am J Gastroenterol. 2007 Aug;102(8):1781-8. doi: 10.1111/j.1572-0241.2007.01279.x. Epub 2007 May 17. PMID 17509029
- [Background] Williams EJ, Taylor S, Fairclough P, Hamlyn A, Logan RF, Martin D, Riley SA, Veitch P, Wilkinson ML, Williamson PR, Lombard M. Risk factors for complication following ERCP; results of a large-scale, prospective multicenter study. Endoscopy. 2007 Sep;39(9):793-801. doi: 10.1055/s-2007-966723. PMID 17703388
- [Background] Wang P, Li ZS, Liu F, Ren X, Lu NH, Fan ZN, Huang Q, Zhang X, He LP, Sun WS, Zhao Q, Shi RH, Tian ZB, Li YQ, Li W, Zhi FC. Risk factors for ERCP-related complications: a prospective multicenter study. Am J Gastroenterol. 2009 Jan;104(1):31-40. doi: 10.1038/ajg.2008.5. PMID 19098846
- [Background] Ding X, Chen M, Huang S, Zhang S, Zou X. Nonsteroidal anti-inflammatory drugs for prevention of post-ERCP pancreatitis: a meta-analysis. Gastrointest Endosc. 2012 Dec;76(6):1152-9. doi: 10.1016/j.gie.2012.08.021. PMID 23164513
- [Background] Elmunzer BJ, Scheiman JM, Lehman GA, Chak A, Mosler P, Higgins PD, Hayward RA, Romagnuolo J, Elta GH, Sherman S, Waljee AK, Repaka A, Atkinson MR, Cote GA, Kwon RS, McHenry L, Piraka CR, Wamsteker EJ, Watkins JL, Korsnes SJ, Schmidt SE, Turner SM, Nicholson S, Fogel EL; U.S. Cooperative for Outcomes Research in Endoscopy (USCORE). A randomized trial of rectal indomethacin to prevent post-ERCP pancreatitis. N Engl J Med. 2012 Apr 12;366(15):1414-22. doi: 10.1056/NEJMoa1111103. PMID 22494121
- [Background] di Sant'Agnese PA, de Mesy Jensen KL, Churukian CJ, Agarwal MM. Human prostatic endocrine-paracrine (APUD) cells. Distributional analysis with a comparison of serotonin and neuron-specific enolase immunoreactivity and silver stains. Arch Pathol Lab Med. 1985 Jul;109(7):607-12. PMID 2409946
- [Background] Elmunzer BJ, Waljee AK, Elta GH, Taylor JR, Fehmi SM, Higgins PD. A meta-analysis of rectal NSAIDs in the prevention of post-ERCP pancreatitis. Gut. 2008 Sep;57(9):1262-7. doi: 10.1136/gut.2007.140756. Epub 2008 Mar 28. PMID 18375470
- [Background] Murray B, Carter R, Imrie C, Evans S, O'Suilleabhain C. Diclofenac reduces the incidence of acute pancreatitis after endoscopic retrograde cholangiopancreatography. Gastroenterology. 2003 Jun;124(7):1786-91. doi: 10.1016/s0016-5085(03)00384-6. PMID 12806612
- [Background] Rome Foundation. Guidelines--Rome III Diagnostic Criteria for Functional Gastrointestinal Disorders. J Gastrointestin Liver Dis. 2006 Sep;15(3):307-12. No abstract available. PMID 17203570
- [Background] Prajapati DN, Hogan WJ. Sphincter of Oddi dysfunction and other functional biliary disorders: evaluation and treatment. Gastroenterol Clin North Am. 2003 Jun;32(2):601-18. doi: 10.1016/s0889-8553(03)00025-6. PMID 12858608
- [Background] Sherman S, Blaut U, Watkins JL, Barnett J, Freeman M, Geenen J, Ryan M, Parker H, Frakes JT, Fogel EL, Silverman WB, Dua KS, Aliperti G, Yakshe P, Uzer M, Jones W, Goff J, Earle D, Temkit M, Lehman GA. Does prophylactic administration of corticosteroid reduce the risk and severity of post-ERCP pancreatitis: a randomized, prospective, multicenter study. Gastrointest Endosc. 2003 Jul;58(1):23-9. doi: 10.1067/mge.2003.307. PMID 12838216
- [Background] Andriulli A, Leandro G, Federici T, Ippolito A, Forlano R, Iacobellis A, Annese V. Prophylactic administration of somatostatin or gabexate does not prevent pancreatitis after ERCP: an updated meta-analysis. Gastrointest Endosc. 2007 Apr;65(4):624-32. doi: 10.1016/j.gie.2006.10.030. PMID 17383459
- [Background] Wu BU, Hwang JQ, Gardner TH, Repas K, Delee R, Yu S, Smith B, Banks PA, Conwell DL. Lactated Ringer's solution reduces systemic inflammation compared with saline in patients with acute pancreatitis. Clin Gastroenterol Hepatol. 2011 Aug;9(8):710-717.e1. doi: 10.1016/j.cgh.2011.04.026. Epub 2011 May 12. PMID 21645639
- [Background] Buxbaum J, Yan A, Yeh K, Lane C, Nguyen N, Laine L. Aggressive hydration with lactated Ringer's solution reduces pancreatitis after endoscopic retrograde cholangiopancreatography. Clin Gastroenterol Hepatol. 2014 Feb;12(2):303-7.e1. doi: 10.1016/j.cgh.2013.07.026. Epub 2013 Aug 3. PMID 23920031
- [Derived] Mok SRS, Ho HC, Shah P, Patel M, Gaughan JP, Elfant AB. Lactated Ringer's solution in combination with rectal indomethacin for prevention of post-ERCP pancreatitis and readmission: a prospective randomized, double-blinded, placebo-controlled trial. Gastrointest Endosc. 2017 May;85(5):1005-1013. doi: 10.1016/j.gie.2016.10.033. Epub 2016 Nov 2. PMID 27816497

RESULTS

PARTICIPANT FLOW:
Groups:
- B (NS+IND): Normal Saline (intravenous during procedure) + Indomethacin (100mg suppository per rectum prior to procedure )
  Indomethacin: Indomethacin is a non-steroidal anti-inflammatory drug (NSAID) which is commonly used to reduce inflammation caused by gout, osteoarthritis and rheumatoid arthritis. It acts by blocking the cyclo-oxygenase 1 and 2 (COX) receptors. It has also been implicated to prevent post-endoscopic retrograde cholangiopancreatography (ERCP) pancreatitis
  Normal Saline: standard IVF would include 0.9% normal saline (NS) solution used during all endoscopic procedures. 0.9% NS includes equal parts sodium and chloride.
Period: Overall Study
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Started | 48 | 48 | 48 | 48
Completed | 48 | 48 | 48 | 48
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND) | Total
Number analyzed (Participants) | 48 | 48 | 48 | 48 | 192
Age, Continuous [Mean (Full Range); unit: years] | 58 [25 to 82] | 62 [19 to 92] | 58 [25 to 91] | 63 [26 to 85] | 60 [19 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 33 | 35 | 23 | 120
  Male | 19 | 15 | 13 | 25 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 1 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 3 | 4 | 13
  White | 32 | 35 | 40 | 40 | 147
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 10 | 8 | 4 | 3 | 25
Region of Enrollment [Number; unit: participants]
  United States | 48 | 48 | 48 | 48 | 192

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Acute Pancreatitis After ERCP as Assessed by Worsening Abdominal Pain Plus Either Elevated Amylase or Lipase 3 x Upper Limit of Normal
Description: amylase or lipase
Time Frame: 30 days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Participants | 10 | 6 | 9 | 3

2. Primary Outcome: The Number of Participants With Acute Pancreatitis After ERCP as Assessed by Worsening Abdominal Pain Plus Imaging Suggestive of Acute Pancreatitis
Description: Imaging may include Computer Tomography
Time Frame: 30 days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Participants | 0 | 1 | 0 | 1

3. Secondary Outcome: The Number of Participants With Acute Respiratory Distress Syndrome (ARDS) After ERCP as Assessed by ARDSnet Criterion (Below)
Description: bilateral opacities on chest imaging not explained by other lung pathology, respiratory failure not explained by heart failure or volume, and overload and a pulmonary arterial oxygen/fraction of inspired oxygen (PaO2/FiO2) ratio under 300, PaO2/FiO2 ratio is the partial pressure arterial oxygen and fraction of inspired oxygen
Time Frame: 30 days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Participants | 1 | 0 | 0 | 0

4. Secondary Outcome: The Number of Participants With Systemic Inflammatory Response Syndrome (SIRS) After ERCP as Assessed by the SIRS Criterion (Below)
Description: Heart rate > 90 beats per minutes
Time Frame: 30 days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Participants | 10 | 6 | 9 | 3

5. Secondary Outcome: The Number of Participants With Systemic Inflammatory Response Syndrome (SIRS) After ERCP as Assessed by the SIRS Criterion (Below)
Description: Respiratory rate > 20 breaths per minute
Time Frame: 30 days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Participants | 10 | 6 | 9 | 3

6. Secondary Outcome: The Number of Participants With Systemic Inflammatory Response Syndrome (SIRS) After ERCP as Assessed by the SIRS Criterion (Below)
Description: PaCO2 < 4.3 kilopascal (kPa) (32 mmHg)
Time Frame: 30 days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Participants | 0 | 0 | 0 | 0

7. Secondary Outcome: The Number of Participants With Systemic Inflammatory Response Syndrome (SIRS) After ERCP as Assessed by the SIRS Criterion (Below)
Description: Temperature < 36°C(96.8°F) or > 38°C(100.4°F)
Time Frame: 30 days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Participants | 10 | 6 | 9 | 3

8. Secondary Outcome: The Number of Participants With Systemic Inflammatory Response Syndrome (SIRS) After ERCP as Assessed by the SIRS Criterion (Below)
Description: white blood cell (WBC) count < 4000 cells/mm³ (4 x 109 cells/L)
Time Frame: 30 days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Participants | 0 | 0 | 0 | 0

9. Secondary Outcome: The Number of Participants With Systemic Inflammatory Response Syndrome (SIRS) After ERCP as Assessed by the SIRS Criterion (Below)
Description: > 10% immature neutrophils (band forms).
Time Frame: 30 days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Participants | 10 | 6 | 9 | 3

10. Secondary Outcome: The Number of Participants With Sepsis After ERCP as Assessed by Infectious Source Defined by Positive Microbiology Culture
Description: positive blood culture
Time Frame: 30 days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Participants | 0 | 0 | 0 | 0

11. Secondary Outcome: The Number of Participants With Multiple Organ Failure (MOF) After ERCP as Assessed by Elevated Creatinine Blood Test
Description: creatinine > 1.5 milligrams/deciliter (mg/dL)
Time Frame: 30 days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Participants | 0 | 1 | 0 | 0

12. Secondary Outcome: The Number of Participants With Multiple Organ Failure (MOF) After ERCP as Assessed by Elevated International Normalized Ratio (INR)
Description: INR > 1.5
Time Frame: 30 days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Participants | 0 | 0 | 0 | 0

13. Secondary Outcome: The Number of Participants With Pancreatic Pseudocyst After ERCP as Assessed by Abdominal Imaging Suggestive of Pseudocyst
Description: Imaging may include Computer Tomography
Time Frame: 30 days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Participants | 0 | 0 | 0 | 1

14. Secondary Outcome: The Number of Participants With Pancreatic Abscess After ERCP as Assessed by Abdominal Imaging Suggestive of Pancreatic Abscess
Description: Imaging may include Computer Tomography
Time Frame: 30 days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Participants | 0 | 0 | 0 | 0

15. Secondary Outcome: The Number of Participants With Perforation After ERCP as Assessed by Abdominal Imaging Suggestive of Perforation
Description: Imaging may include Computer Tomography
Time Frame: 30 days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Participants | 0 | 0 | 0 | 0

16. Secondary Outcome: The Number of Participants Who Undergo Surgery After ERCP, as Assessed by Surgical Operative Report
Time Frame: 30 days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Participants | 0 | 0 | 0 | 0

17. Secondary Outcome: The Number of Participants With Mortality After ERCP as Assessed by Medical Record Reporting
Time Frame: 30 days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Participants | 1 | 2 | 2 | 1

18. Secondary Outcome: The Number of Participants With Post-procedural Medical Care (ED Visit, Urgent Care, Hospitalization) as Assessed by Medical Record and Patients Self-reporting
Time Frame: 30 days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Participants | 6 | 2 | 2 | 1

19. Secondary Outcome: The Length of Stay (LOS) of Participants After ERCP if Medical Care is Sought as Assessed in Days
Time Frame: 30 days after ERCP
Measure: Mean (Standard Deviation); unit: days
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
days | 2.3 (3.5) | 2.2 (4.1) | 1.9 (3.4) | 4.3 (8.4)

20. Secondary Outcome: The Number of Participants Who Were Readmitted After ERCP as Assessed by Medical Record and Patients Self-reporting
Time Frame: 30 days after ERCP
Measure: Count of Participants; unit: Participants
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Participants | 6 | 2 | 2 | 1
Statistical Analysis 1: Comparison: A (NS+Placebo) vs D (LR+IND); Test type: Superiority; p = 0.04, Fisher Exact

ADVERSE EVENTS:
Time Frame: 30 days
Description: In the case of delayed adverse events (AE), all patients were encouraged to return to the institution in which their procedure was performed. To ensure comprehensive data collection, participants received a telephone call or in person encounter (when hospitalized) within 24 hours and also at 30 days from their procedure
Arm/Group | A (NS+Placebo) | B (NS+IND) | C (LR+Placebo) | D (LR+IND)
All-Cause Mortality (participants affected / at risk) | 1/48 | 2/48 | 2/48 | 1/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48 | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 2/48 | 1/48 | 1/48 | 1/48
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A (NS+Placebo) (N=48) | B (NS+IND) (N=48) | C (LR+Placebo) (N=48) | D (LR+IND) (N=48)
Acute Renal Failure (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — Acute renal failure defined as creatinine > 1.2 mg/dL
Pulmonary Edema (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splenic Laceration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
We did not power this study to detect a difference between our other comparative groups (NS+IND, LR+placebo), these comparisons may have been prone to type II statistical errors. Single center experience is another possible limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes